CLINICAL TRIAL: NCT04607681
Title: Evaluation of the Effect of Web-designed Training Developed for Asthma Patients on Drug Compliance, Asthma Control, and Fatigue
Brief Title: Evaluation of the Effect of Web-designed Training Developed for Asthma Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eskisehir Osmangazi University (Other)
Responsible Party: Principal Investigator, EYLUL GULNUR ERDOGAN, Phd, PHD STUDENT, Eskisehir Osmangazi University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: Eskisehir Osmangazi Universty
Record Dates: First submitted 2020-10-20; First posted 2020-10-29 (Actual); Last update posted 2022-09-19 (Actual); Status verified 2022-09

CONDITIONS: Asthma
Keywords: asthma; compliance; life quality; asthma control; web based training; asthma education
MeSH Terms: conditions — Asthma; Patient Compliance | interventions — Educational Status

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 1 GROUP (Experimental): Patients who agree to participate in the study will be informed about the study and their written and verbal consent will be obtained. At this stage, which will last 6 weeks for each patient;
  * On the first day, the patients will be evaluated first by filling the "Individual Descriptive Features Form, Information Need Determination Question Form, COPD and Asthma Fatigue Scale, Medication Compliance Notification Scale, Asthma Control Test (ACT), Form for evaluation of the skills of using inhalation devices",
  * In order for the patients in the intervention group to use the web-based asthma education program, a web-based asthma education program will be introduced by giving their username and password.
  After 6 weeks of training, second data will be collected on the web in the intervention group.
  Interventions: Behavioral: EDUCATION
- 2 GROUP (No Intervention): Written and verbal consents will be obtained from patients who agree to participate in the study by providing information about the study.
  At this stage, which will take 6 weeks for each patient; On the first day, the patients will first be evaluated by filling the "Individual Descriptive Characteristics Form, Information Requirement Determination Question Form, COPD and Asthma Fatigue Scale, Medication Compliance Notification Scale, Asthma Control Test (ACT), Form for evaluation of the skills of using inhalation devices", Second data after 6 weeks will be collected in the control group via Google form or phone call

INTERVENTIONS:
Behavioral: EDUCATION — WEB BASED EDUCATION
  Arms: 1 GROUP

SUMMARY:
The study is an experimental study with pre-test-post-test control group in order to determine the effect of web-designed training developed for asthma patients on drug compliance, asthma control, and fatigue

DETAILED DESCRIPTION:
In the first stage, it is aimed to develop, implement and evaluate a web designed asthma education program for asthma patients. In the second stage, it is to evaluate the effect of the web-designed education program developed for asthmatic patients on drug ompliance, asthma control, and fatigue The population of the study consists of patients diagnosed with asthma who are registered in Family Health Centers in Eskişehir. The individuals that constitute the target group in the study will be determined through the records of patients diagnosed with asthma registered in the family health center or the list of patients in the J45-Asthma and J46 Status Asthmaticus ICD codes. The sample of the study will be the patients who meet the criteria for inclusion in the study. G power analysis program was used to determine the sample size. The research will be conducted in two groups, an intervention and a control group. The sample size of the research was found to be 200.

In collecting research data; The personal descriptive characteristics form prepared by the researcher, the questionnaire for determining the information needs, Form for evaluation of the skills of using inhalation devices and the opinion form regarding the web-based asthma education program will be used. At the same time, COPD and asthma fatigue scale, drug compliance reporting scale and Asthma Control Test (AKT) will be used.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and over,
* Those who have been diagnosed with asthma for at least one year
* Those with poor asthma control
* Using at least one asthma medication
* Not having a communication problem, such as inability to understand/speak Turkish, that would prevent participating in the research or receiving training,
* Being literate,
* Having an internet connection at home or on their phone,
* Having and using a computer, tablet or smart phone,
* Patients who accepted to participate in the study voluntarily formed the sample of the study.

Exclusion Criteria:

* No internet connection at home or on their phone,
* Do not know how to use the Internet and computer,
* Having a communication problem, such as inability to understand/speak Turkish, that would prevent participating in the research or receiving training,
* Illiterate,
* Diagnosed with another respiratory system disease,
* Diagnosed with cancer or undergoing cancer treatment,
* Those who have been diagnosed with or have had COVID-19,
* Individuals with a psychiatric illness were not included in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2021-07-21 (Actual); Primary Completion 2021-11-10 (Actual); Study Completion 2022-01-24 (Actual)

PRIMARY OUTCOMES:
change from baseline in Medication Compliance Reporting Scaleat week 6 | baseline and 6 weeks
  Medication Compliance Reporting Scale Participants are asked to indicate the frequency of the 5 statements in each of them.
  The scale is evaluated with a 5-point Likert type such that 5 = never, 4 = rarely, 3 = sometimes, 2 = often and 1 = always.
  The total test score is obtained by summing the scores obtained from the items. The scores obtained from the scale range from 5 to 25. An increase in the obtained scores indicates compatibility, and a decrease in scores indicates incompatibility.
change from baseline in COPD and Asthma Fatigue Scale (DAS) at week 6 | baseline and 6 weeks
  COPD and Asthma Fatigue Scale (DAS) The scale consists of 12 items, and a Likert type rating (1 = never, 2 = rarely, 3 = sometimes, 4 = often, 5 = very often) is used for its answers.
  In calculating the scale score, the first 10 questions correspond to never = 1 point, rarely = 2 points, sometimes = 3 points, often = 4 points, very often = 5 points, and in the 11th and 12th questions never = 5 points, rarely = 4 points. , sometimes = 3 points, often = 2 points, very often = 1.
  The total raw score is determined by adding the scores of each item and the raw scores are converted into a total scale score between 0-100. The higher the score obtained from the scale indicates that the fatigue level of the person is high.
change from baseline in Asthma Control Test (AKT) at week 6 | baseline and 6 weeks
  Asthma Control Test (AKT); This scale consists of five Likert type and consists of five questions.
  The maximum score of this test is 25 and the minimum score is 5, while 25 points are "full control", 20-24 points "good control" and a score of less than 19 is considered "uncontrolled"
change from baseline in bility to use inhalation devices at week 6 | baseline and 6 weeks
  Form for evaluation of the skills of using inhalation devices
evaluating the web-based asthma education program | at 6 weeks
  Opinion Form Regarding the Web Based Asthma Education Program
  This form contains 20 questions prepared to determine the views of asthma patients on the web-based asthma education program.

CONTACTS AND LOCATIONS:
Overall Officials: Ozlem Orsal, Prof, Study Director — Eskisehir Osmangazi University
Locations (1):
- Eskisehir Osmangazi Universty, Eskişehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Schatz M, Sorkness CA, Li JT, Marcus P, Murray JJ, Nathan RA, Kosinski M, Pendergraft TB, Jhingran P. Asthma Control Test: reliability, validity, and responsiveness in patients not previously followed by asthma specialists. J Allergy Clin Immunol. 2006 Mar;117(3):549-56. doi: 10.1016/j.jaci.2006.01.011. PMID 16522452
- [Background] Schatz M, Zeiger RS, Drane A, Harden K, Cibildak A, Oosterman JE, Kosinski M. Reliability and predictive validity of the Asthma Control Test administered by telephone calls using speech recognition technology. J Allergy Clin Immunol. 2007 Feb;119(2):336-43. doi: 10.1016/j.jaci.2006.08.042. Epub 2006 Dec 27. PMID 17194469
- [Background] Koufopoulos JT, Conner MT, Gardner PH, Kellar I. A Web-Based and Mobile Health Social Support Intervention to Promote Adherence to Inhaled Asthma Medications: Randomized Controlled Trial. J Med Internet Res. 2016 Jun 13;18(6):e122. doi: 10.2196/jmir.4963. PMID 27298211